CLINICAL TRIAL: NCT04217213
Title: Effect of Intercostal Nerve Block With Ropivacaine Combined With Mecobalamine on Chronic Pain After Thoracic Surgery -- a Single-center Randomized, Double-blind Controlled Trial
Brief Title: Effect of Intercostal Nerve Block With Ropivacaine Combined With Mecobalamine on Chronic Pain After Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Han Yuan, associate chief physician, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XYFY2019-KL169-01
Record Dates: First submitted 2019-11-30; First posted 2020-01-03 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ropivacaine combined with mecobalamine (Experimental): Intercostal nerve block with 0.5% ropivacaine combined with mecobalamine (0.5mg).
  Interventions: Procedure: Intercostal nerve block
- ropivacaine (Active Comparator): Intercostal nerve block with 0.5% ropivacaine alone.
  Interventions: Procedure: Intercostal nerve block

INTERVENTIONS:
Procedure: Intercostal nerve block — In the experimental group, the surgeons used 0.5% ropivacaine combined with mecobalamine (0.5mg) before the operation to perform intercostal nerve block in the operating incision, closed thoracic drainage incision and one intercostal nerve block in each upper and lower costal cavity, and injected 5ml in each intercostal nerve block.In the control group, surgeons used 0.5% ropivacaine alone before the operation to perform intercostal nerve block through the operating incision, closed thoracic drainage incision and one intercostal nerve block in each upper and lower costal cavity. 5ml was injected into each intercostal nerve block.

SUMMARY:
This project intends to investigate the effects of intercostal nerve block with ropivacaine combined with mecobalamin on chronic post-surgical pain (CPSP) in thoracic postoperative patients. Related clinical characteristics of postoperative chronic pain. The results of the study provide clinicians with a simple and inexpensive new method of preventing CPSP, in order to prevent the occurrence of CPSP and reduce the incidence of CPSP, thereby reducing CPSP to patients and their families, hospitals. And public resources.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, conscious;
2. ASA class Ⅰ ~ Ⅲ;
3. Thoracoscopic lobectomy was proposed;
4. The han nationality;
5. Native speaker of Chinese;
6. Agree to participate in this study and sign the informed consent.

Exclusion Criteria:

1. Patients allergic to meccobalamin or ropivacaine;
2. Patients with previous history of chest surgery;
3. Patients with tumor invasion of chest wall, abscess, tumor intercostal neuropathy or pathological rib fracture;
4. Patients with a history of analgesic addiction or abuse, epilepsy, one or other neurological disease;
5. Diabetic patients;
6. Patients who need other drugs for pain relief but have not completed treatment or have completed treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of chronic pain after chest surgery | At the 3rd month after surgery
  The incidence of chronic pain after chest surgery was measured by NRS(numeric rating scales) at the 3rd month after surgery.For pain evaluation,we used the 11 point numeric rating scale(NRS),where an NRS scores of 0 represented "no pain" and a score of 10 represented "worst pain imaginable".

SECONDARY OUTCOMES:
The incidence of acute pain after chest surgery | 24 to 72 hours after surgery
  An NRS score was performed 24 to 72 hours after surgery to determine the incidence of acute pain after thoracic surgery.For pain evaluation,we used the 11 point numeric rating scale(NRS),where an NRS scores of 0 represented "no pain" and a score of 10 represented "worst pain imaginable".
Incidence of postoperative neuropathic pain | At the 3rd month after surgery
  The incidence of neuropathic pain was measured by DN4 scale at the 3rd month after surgery.Douleur Neuropathique 4 (DN4) is a screening questionnaire to help identify neuropathic pain (NP) in clinical practice and research,where a DN4 scores greater than or equal to 4 represented the patients had "postoperative neuropathic pain".
Incidence of other postoperative complications | At the 3rd month after surgery
  Postoperative complications included that pulmonary complications, delirium, intestinal obstruction, pulmonary embolism, acute respiratory failure, acute renal failure, incision infection, cerebrovascular accident and other complications related to surgery.
Incidence of readmission within 30 days after surgery | At the 30 days after surgery
  The incidence and the reason of readmission within 30 days after surgery was obtained through postoperative follow-up.
Incidence of death within 30 days after surgery | At the 30 days after surgery
  The incidence and the reason of death within 30 days after surgery was obtained through postoperative follow-up
Length of stay | At the 3rd month after surgery
  The total length of hospital stay.
Cost of stay | At the 3rd month after surgery
  The total cost of hospital stay.
icu length of stay | At the 3rd month after surgery
  The number of hours of postoperative stay in ICU.
Incidence of secondary operation | At the 3rd month after surgery
  Whether the patient has a second operation and the reason and the incidence of this operation.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology of the Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China